CLINICAL TRIAL: NCT07272460
Title: Time Restricted-eating and Metabolic Health in Patients With Type 2 Diabetes
Brief Title: Time Restricted-EAting for Type 2 Diabetes and MEtabolic Health: the TEA TIME Trial
Acronym: TEA-TIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB # 0002
Record Dates: First submitted 2025-09-29; First posted 2025-12-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Overweight (BMI > 25)
Keywords: Randomized controlled trial; Time-restricted eating; Intermittent fasting; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (Experimental): Time-restricted eating protocol consisting of time-restricted eating with 18 hours of fasting and 6 hour window of eating (between 2 to 8 PM) every day.
  Interventions: Behavioral: Time-restricted eating
- Standard lifestyle (Active Comparator): Standard lifestyle recommendation as per Diabetes Canada Guidelines.
  Interventions: Behavioral: Standard lifestyle

INTERVENTIONS:
Behavioral: Time-restricted eating — 18 hours of fasting and 6 hour window of eating (between 2 to 8 PM) every day for 52 weeks.
  Arms: Time-restricted eating
Behavioral: Standard lifestyle — standard lifestyle recommendations as per Diabetes Canada guidelines [where patients are encouraged to maintain regularity in timing and spacing of meals with no specific recommendation regarding hours of fasting]
  Arms: Standard lifestyle

SUMMARY:
Time-restricted eating - where no food is consumed over a period of time - has been shown to promote weight loss and improve cardio-metabolic function. In individuals with type 2 diabetes, it is also been shown to improve glucose control. The investigators propose a randomized controlled trial to determine whether time-restricted eating is an effective therapeutic strategy that can preserve pancreatic beta-cell function and improve glycemic control early in participants with type 2 diabetes.

DETAILED DESCRIPTION:
In this study, eligible patients with type 2 diabetes will be randomized to either time-restricted eating or standard lifestyle. The hypothesis under study is whether time-restricted eating can improve pancreatic beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with previously diagnosed BMI ≥ 25 kg/m2 and type 2 diabetes within preceding 10 years.
* Age 18 - 75 years inclusive
* Stable weight over past 12 weeks (less than 5% change in body weight) (self-reported)
* Diabetes treatment consisting of lifestyle only or metformin, dipeptidyl peptidase-4 (DPP-4) inhibitor, and sodium-glucose co-transporter 2 (SGLT2) inhibitors either as monotherapy or in combination.
* Ability to read and understand English

Exclusion Criteria:

* Current diabetes treatment with insulin, glucagon-like peptide-1 receptor agonists, and/or sulfonylureas.
* Use of any other pharmacological treatment for weight-loss
* Previous surgical treatment for weight loss such as gastric bypass or gastric band
* Any history of eating disorder
* Currently pregnant or lactating
* Renal dysfunction as evidenced by estimated glomerular filtration rate < 25 ml/min by CKD-EPI Creatinine Equation
* New York Heart Association class II-IV heart failure
* Hepatic disease considered to be clinically significant (includes jaundice, chronic hepatitis, or previous liver transplant) or transaminases >2.5X the upper limit of normal
* Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer)
* Any other factor likely to limit adherence to the study, in the opinion of the investigators
* Concurrent participation in another research study relevant to diabetes and metabolic health

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Differences in baseline-adjusted Insulin-Secretion-Sensitivity Index-2 (ISSI-2) between the study groups. | 52-weeks
  Baseline-adjusted beta-cell function at 52 weeks, measured by Insulin Secretion-Sensitivity Index-2 (ISSI-2).

SECONDARY OUTCOMES:
Differences in baseline-adjusted insulin resistance between the study groups | 52-weeks
  Baseline-adjusted insulin resistance at 52-weeks measured by HOMA-IR
Differences in time in glucose target range between each study group | 52-weeks
  Time in glucose target range indicates the amount of time (in %) that glucose readings are within the defined target glucose range of 3.9-10.0 mmol/L.

OTHER OUTCOMES:
Anthropometric measures | 52-weeks
  Differences in body weight (kg) between each study arm
Additional measures of beta-cell function | 52-weeks
  Insulinogenic index/HOMA-IR.
Additional measures of insulin sensitivity | 52-weeks
  Matsuda Index
Time above glucose target on isCGM | 52 weeks
  Differences between each study arm in time-above target of 10 mmol/l (%) obtained by isCGM (FreeStyle Libre devices).
Additional anthropometric measures | 52 weeks
  Differences in waist circumference between the study arms

CONTACTS AND LOCATIONS:
Locations (1):
- Leadership Sinai Centre for Diabetes, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No